CLINICAL TRIAL: NCT01421914
Title: Determining the Minimum Effective Volume of Local Anesthetic for Ultrasound-guided Axillary Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, MD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Unifesp-USG Axillary block
Record Dates: First submitted 2011-08-21; First posted 2011-08-23 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Axillary Brachial Plexus Block
Keywords: Ultrasound; Axillary block; Bupivacaine; Minimum; Volume; Minimum volume of bupivacaine 0,5%

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bupivacaine 0,5% (Other): Single arm study
  Interventions: Other: Bupivacaine 0,5%

INTERVENTIONS:
Other: Bupivacaine 0,5% — The study method was a step-up/step-down sequence model where the dose for following patients was determined by the outcome of the preceding block. The starting dose of bupivacaine was 5 mL per nerve. In the case of block failure, the dose was increased by 0.5 mL per nerve. Conversely, block success resulted in a reduction in dose by 0.5 mL per nerve. Each of the three nerves was treated as a separate entity. Dose adjustments were made to each nerve individually. The volume dose was increased in 0.5 mL at every 5 consecutive cases regardless of the result of the previous block in order to minimize bias occurence. A blinded assistant assessed sensory and motor blockade at 5-min intervals up to 30 min.

SUMMARY:
This is a study to calculate the minimum effective volume of bupivacaine 0,5% with epinephrine for successful axillary brachial plexus block for hand surgery in 50% of the patients (MEV50).

DETAILED DESCRIPTION:
Study Design All patients had their demographic data recorded upon inclusion in the study. Routine preoperative monitoring was subsequently performed using ECG, non-invasive blood pressure measurements and pulse oximetry. Intravenous access was established and maintained with a crystalloid infusion.

The axillary approach using ultrasound (M-Turbo ® System with HFL 38x linear transducer 13-6 MHz, SonoSite, Bothell, WA, USA) and peripheral nerve stimulation (Stimuplex ® DIG RC, B. Braun, Melsung, Germany) guidance was performed to obtain brachial plexus block with the patient lying in the supine position. The needle used was a 22G x 50 mm (AEQ2250, BMD Group, Venezia, Italy). The puncture site was infiltrated with lidocaine 1% after asepsis and antisepsis skin treatment with chlorhexidine. After that, the ulnar, radial, median and musculocutaneous nerves were visualized by ultrasound (Figure 1) and had their identity confirmed by nerve stimulation. An initial dose of 5 mL of bupivacaine 0.5% with adrenaline (1:200,000) was injected in the proximity of each nerve. If severe pain at the injection was referred or, if nerve diameter changed during injection, injection was immediately interrupted, patient was removed form study and followed postoperatively for possible intraneural injection. The needle was repositioned during injection and perineural injected was ensured by ultrasound.

The efficacy of the block was assessed by an assessor blinded to injected volume. Assessments were conducted every 5 min up to a total of 30 min following the end of the injection of the local anaesthetic. Block assessment was finished either after surgical anaesthesia was achieved or,after 30 min had elapsed.

Success or failure of the block was used to dynamically reduce or increase, respectively, the volume of local anaesthetic that was used for the subsequent patient. When a block was achieved, the subsequent patient received a 0.5 mL reduction in the total volume of local anaesthetic per nerve. Upon failure of the block, the patient received a complementation of nerve blocks at a point distal to the axilla, and the volume of local anaesthetic delivered to the next patient was increased by 0.5 mL. After the block was assessed, the patients were cleared for surgery. During surgery, an infusion of 25-50 mcg.kg-1.min-1 of propofol was used to achieve proper sedation. Also, if during the procedure pain was referred, the block was considered failure and a conversion to general anaesthesia was performed.

After surgery, the patients were admitted to the post-anaesthetic recovery room, where they were continuously monitored using ECG as well as non-invasive blood pressure and pulse oximetry until the requirements for discharge were met. Postoperative analgesia was evaluated in the recovery room using a visual analogue pain scale (VAS) three hours after the block.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 adult patients scheduled for ambulatorial hand surgery were included

Exclusion Criteria:

* cognitive impairment,
* coagulopathy,
* allergy to bupivacaine,
* infection at the puncture site,
* body mass index > 35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Determining the minimum effective volume of bupivacaine 0,5% with epinephrine For successful axillary brachial plexus block for hand surgery | A blinded Assistant assess sensory and motor blockade in a 5-min intervals up to 30 minutes.
  Assessment of the success of ABPB A motor function score of 2 or less on the modified Bromage scale and also a lack of thermal sensitivity and response to a pinprick in the regions of the median, ulnar, radial and musculocutaneous nerves were considered characteristics of a successful block. Moreover, the surgery should be concluded without any complementary analgesia to confirm the success of the anaesthetic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil